CLINICAL TRIAL: NCT01413581
Title: A Prospective, Randomized, Double-Blind, Phase 3 Study Comparing rhBSSL and Placebo Added to Infant Formula or Pasteurized Breast Milk During 4 Weeks of Treatment in Preterm Infants Born Before Week 32 of Gestational Age
Brief Title: Comparison of rhBSSL With Placebo When Added to Infant Formula or Pasteurized Breast Milk During 4 Weeks of Treatment in Preterm Infants
Acronym: LAIF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary endpoint showed no stat significant difference. FU > M12 terminated.
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BVT.BSSL-030
Record Dates: First submitted 2011-06-08; First posted 2011-08-10 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Prevention of Growth Restriction
Keywords: rhBSSL; preterm infants; Swedish Orphan Biovitrum; growth velocity; Prevention of growth restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBSSL (Experimental): rhBSSL (recombinant human bile-salt-stimulated lipase)
  Interventions: Drug: rhBSSL (recombinant human bile-salt-stimulated lipase)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhBSSL (recombinant human bile-salt-stimulated lipase) — rhBSSL added to infant formula/pasteurized breast milk during a 4 week treatment period.
  Arms: rhBSSL
Drug: Placebo — Placebo added to infant formula/pasteurized breast milk during a 4 week treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that rhBSSL improves growth in preterm infants as compared with placebo.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that rhBSSL improves growth in preterm infants as compared with placebo. The infants should be born before week 32 of gestational age.

The study drug, rhBSSL or placebo, will be administered during a 4 week treatment period by adding it to either infant formula or pasteurized breast milk.

The study will also evaluate the safety and tolerability of rhBSSL.

Eligible patients will be randomized in a ratio of 1:1 (rhBSSL:placebo). The study consists of maximum 1 week screening period, a 4-week treatment period and a 2 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born before week 32 of gestation.
* Preterm infant who is less than 33 weeks postmenstrual age at the time of randomization.
* Preterm infant who is appropriate for gestational age (AGA) or small for gestational age (SGA) at birth.
* Preterm infant who is receiving food enterally (bottle or gavage tube) at a level of at least 100 ml/kg/day at randomization.
* Preterm infant whose enteral feeding consists of only infant formula or only pasteurized breast milk at the time of inclusion, and who are expected to remain on only infant formula for 4 weeks, or only pasteurized breast milk for at least 2 weeks following treatment initiation.
* Preterm infant who is expected not to receive any fresh breast milk for 4 weeks following treatment initiation.
* Informed consent is obtained.

Exclusion Criteria:

* Expected stay in the hospital is less than 4 weeks from the first dose of study drug.
* Criteria to ensure no disease or treatment affecting growth or development, e.g. brain disease, necrotizing enterocolitis.
* Enrolled in another concurrent clinical intervention study.

Max Age: 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 415 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Growth velocity in grams per kilogram per day during 4 weeks of treatment. | Baseline and Day 29

SECONDARY OUTCOMES:
Change from baseline in body weight (g) at 3 months | Baseline and Month 3
Body weight (g) at 12 months' corrected age | 12 months´ corrected age
Body weight (g) at 24 months' corrected age | 24 months´ corrected age
Change from baseline in total body length (mm) at 4 weeks | Baseline and Day 29
Change from baseline in total body length (mm) at 3 months | Baseline and Month 3
Total body length (mm) at 12 months' corrected age | 12 months' corrected age
Total body height (cm) at 24 months' corrected age | 24 months' corrected age
Growth restriction | Day 29
  Defined as growth velocity <15 gram per kilogram bodyweight per day during 4 weeks of treatment
Time to readiness for discharge | Baseline and date of readiness for discharge
  Time until each of the following are fulfilled
  * sustained weight gain (weight of 1800 g sustained for three days)
  * ability to maintain normal body temperature
  * ability to suckle feed
  * ability to maintain stable cardiorespiratory function
Time to discharge | Baseline and date of discharge
Change from baseline in head circumference (mm) at 4 weeks. | Baseline and Day 29
Change from baseline in head circumference (mm) at 3 months. | Baseline and Month 3
Head circumference (mm) at 12 months' corrected age. | 12 months´ corrected age
Head circumference (mm) at 24 months' corrected age. | 24 months´ corrected age
Time from baseline to 150 mL/kg/day of enteral feeding | Date of first dose and date 150 mL/kg/day of enteral feeding achieved (or exceeded)
Re-admission to hospital within 1 month of discharge | Date of discharge and date of re-admission
Bayley Scale of Infant and Toddler Development, third edition: Cognitive domain composite score 12 months' corrected age | 12 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Cognitive domain composite score at 24 months' corrected age | 24 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Language domain composite score at 12 months' corrected age | 12 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Language domain composite score at 24 months' corrected age | 24 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Motor domain composite score at 12 months' corrected age | 12 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Motor domain composite score at 24 months' corrected age | 24 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Social-emotional domain composite score at 24 months' corrected age | 24 months' corrected age
Bayley Scale of Infant and Toddler Development, third edition: Adaptive behavior domain composite score at 24 months' corrected age | 24 months' corrected age
Neurodevelopment Disability Composite | 24 months' corrected age
  Presence of :
  * Composite score of less than 70 on any of the cognitive, language or motor domains of Bayley scale of infant and toddler development, third edition
  * Bilateral deafness
  * Bilateral blindness
  * Cerebral palsy
Child Behavior Checklist total problem score at 24 months' corrected age | 24 months' corrected age visit
Number of patients with at least one treatment emergent Adverse Event | Baseline and Day 29
  Total and by system organ class and preferred term (coded by MedDRA)
Number of patients with at least one treatment emergent Adverse Event | Day 29 and Month 3
  Total and by system organ class and preferred term (coded by MedDRA)
Number of patients with at least one treatment emergent Serious Adverse Event | Baseline and Day 29
  Total and by system organ class and preferred term (coded by MedDRA)
Number of patients with at least one treatment emergent Serious Adverse Event | Day 29 and Month 3
  Total and by system organ class and preferred term (coded by MedDRA)
Number of patients with at least one Serious Adverse Drug Reaction | 12 months' corrected age and 24 months' corrected age
  Total and by system organ class and preferred term (coded by MedDRA)
Level of Vitamin A (nmol/L) at 4 weeks | Day 29
Level of Vitamin D (nmol/L) at 4 weeks | Day 29
Number of outpatient visits from the time of initial hospital discharge to home up to 24 months' corrected age | Date of initial hospital discharge to home to date of 24 months' corrected age
Number of inpatient visits from the time of initial hospital discharge to home up to 24 months' corrected age | Date of initial hospital discharge to home to date of 24 months' corrected age
Number of days of hospitalization from the time of initial hospital discharge to home up to 24 months' corrected age | Date of initial hospital discharge to home to date of 24 months' corrected age
Number of days in intensive care unit from the time of initial hospital discharge to home up to 24 months' corrected age | Date of initial hospital discharge to home to date of 24 months' corrected age
Number of days lost from work related to the child's condition from the time of initial hospital discharge to home up to 24 months' corrected age | Date of initial hospital discharge to home to date of 24 months' corrected age
Presence of chronic medical conditions/diagnoses at 24 months' corrected age | 24 months' corrected age
Docosahexaenoic acid (% of total fatty acids) in the serum triglyceride fraction at 4 weeks | Day 29
Docosahexaenoic acid (% of total fatty acids) in the serum phosphatidylcholine fraction at 4 weeks | Day 29
Arachidonic acid (% of total fatty acids) in the serum triglyceride fraction at 4 weeks | Day 29
Arachidonic acid (% of total fatty acids) in the serum phosphatidylcholine fraction at 4 weeks | Day 29
Number of patients with antibodies to rhBSSL at 4 weeks | Day 29
Number of patients with antibodies to rhBSSL at Month 3 | Month 3
Number of patients with antibodies to rhBSSL at 12 months' corrected age | 12 months' corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Timdahl, MD, Study Director — Swedish Orphan Biovitrum
Locations (49):
- Belgium (5):
  - Swedish Orphan Biovitrum Investigational Site, Bruges
  - Swedish Orphan Biovitrum Investigational Site, Leuven
  - Swedish Orphan Biovitrum Investigational Site, Liège
  - Swedish Orphan Biovitrum Investigational Site, Rocourt
  - Swedish Orphan Biovitrum Investigational Site, Wilrijk
- Czechia (4):
  - Swedish Orphan Biovitrum Investigational Site, Hradec Králové
  - Swedish Orphan Biovitrum Investigational Site, Olomouc
  - Swedish Orphan Biovitrum Investigational Site, Prague
  - Swedish Orphan Biovitrum Investigational Site, Zlín
- France (7):
  - Swedish Orphan Biovitrum Investigational Site, Amiens
  - Swedish Orphan Biovitrum Investigational Site, Lille
  - Swedish Orphan Biovitrum Investigational Site, Nancy
  - Swedish Orphan Biovitrum Investigational Site, Paris
  - Swedish Orphan Biovitrum Investigational Site, Rouen
  - Swedish Orphan Biovitrum Investigational Site, Strasbourg
  - Swedish Orphan Biovitrum Investigational Site, Toulouse
- Germany (4):
  - Swedish Orphan Biovitrum Investigational Site, Berlin
  - Swedish Orphan Biovitrum Investigational Site, Freiburg im Breisgau
  - Swedish Orphan Biovitrum Investigational Site, Heidelberg
  - Swedish Orphan Biovitrum Investigational Site, Wiesbaden
- Hungary (6):
  - Swedish Orphan Biovitrum Investigational Site, Budapest
  - Swedish Orphan Biovitrum Investigational Site, Gyula
  - Swedish Orphan Biovitrum Investigational Site, Miskolc
  - Swedish Orphan Biovitrum Investigational Site, Nyíregyháza
  - Swedish Orphan Biovitrum Investigational Site, Pécs
  - Swedish Orphan Biovitrum Investigational Site, Veszprém
- Italy (6):
  - Swedish Orphan Biovitrum Investigational Site, Ancona
  - Swedish Orphan Biovitrum Investigational Site, Bari
  - Swedish Orphan Biovitrum Investigational Site, Foggia
  - Swedish Orphan Biovitrum Investigational Site, Milan
  - Swedish Orphan Biovitrum Investigational Site, Padua
  - Swedish Orphan Biovitrum Investigational Site, Roma
- Poland (5):
  - Swedish Orphan Biovitrum Investigational Site, Bydgoszcz
  - Swedish Orphan Biovitrum Investigational Site, Gdansk
  - Swedish Orphan Biovitrum Investigational Site, Lodz
  - Swedish Orphan Biovitrum Investigational Site, Poznan
  - Swedish Orphan Biovitrum Investigational Site, Warsaw
- Russia (2):
  - Swedish Orphan Biovitrum Investigational Site, Ivanovo
  - Swedish Orphan Biovitrum Investigational Site, Nizhny Novgorod
- Spain (8):
  - Swedish Orphan Biovitrum Investigational Site, Almería
  - Swedish Orphan Biovitrum Investigational Site, Cadiz
  - Swedish Orphan Biovitrum Investigational Site, Córdoba
  - Swedish Orphan Biovitrum Investigational Site, Madrid
  - Swedish Orphan Biovitrum Investigational Site, Málaga
  - Swedish Orphan Biovitrum Investigational Site, Oviedo
  - Swedish Orphan Biovitrum Investigational Site, Salamanca
  - Swedish Orphan Biovitrum Investigational Site, Santiago de Compostela
- Sweden (2):
  - Swedish Orphan Biovitrum Investigational Site, Stockholm
  - Swedish Orphan Biovitrum Investigational Site, Umeå

REFERENCES:
- [Derived] Casper C, Hascoet JM, Ertl T, Gadzinowski JS, Carnielli V, Rigo J, Lapillonne A, Couce ML, Vagero M, Palmgren I, Timdahl K, Hernell O. Recombinant Bile Salt-Stimulated Lipase in Preterm Infant Feeding: A Randomized Phase 3 Study. PLoS One. 2016 May 31;11(5):e0156071. doi: 10.1371/journal.pone.0156071. eCollection 2016. PMID 27244221
- [Derived] Casper C, Carnielli VP, Hascoet JM, Lapillonne A, Maggio L, Timdahl K, Olsson B, Vagero M, Hernell O. rhBSSL improves growth and LCPUFA absorption in preterm infants fed formula or pasteurized breast milk. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):61-9. doi: 10.1097/MPG.0000000000000365. PMID 25222806
- See also: Results are available on the European Union Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2010-023909-35/results